CLINICAL TRIAL: NCT01835717
Title: Cross-sectional Study for Cognitive and Genetic Characterization of a 45-65 Years Old Population
Brief Title: Study for Cognitive and Genetic Characterization of a 45-65 Years Old Population
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Obra Social La Caixa, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: Study 45-65/FPM 2012
Record Dates: First submitted 2013-04-15; First posted 2013-04-19 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Healthy Individuals
Keywords: Preclinical phase of Alzheimer's disease; Asymptomatic phase of Alzheimer's disease; Cognitive normal; Exogenous factors; Endogenous factors; Episodic memory test; Executive function test; Memory binding test validation into Spanish; Memory binding test validation into Catalan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum; white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cognitively normal individuals

SUMMARY:
Before Alzheimer's disease (AD) clinical symptoms appear, there is a long period when changes in the brain occur. In this long asymptomatic period or preclinical phase, studies with populations at risk of developing AD have shown cognitive differences compared to control groups without such risk. There is a need for short, sensitive, easily administered, reproducible, non-expensive and independent of socio-demographic influences tests enabling the detection of pre-symptomatic variations in memory, when the memory decline is still within a normal range.

Study main hypothesis: When evaluated with high-demanding tests of memory and executive function, the cognitive performance of cognitive healthy people aged between 45 and 65 and, extensively, to a group of up to 75 years, will vary significantly depending on clinical, socio-demographic and genetic features

DETAILED DESCRIPTION:
The purpose of Study 45-65 is to assess if:

* Endogenous factors (clinical history, risk factors, genetic factors APOE4, etc…), exogenous (socio-demographic, ambient and lifestyle variables) and cognitive reserve (including bilingualism) influence cognitive performance.
* New and/or updated tests translated and validated in Spanish and Catalan when needed, will provide accurate and sensitive measurements of the variability of cognitive performance in this target population, representative of the preclinical phase of Alzheimer's disease.

An optional visit is offered to study participants that includes: cerebral magnetic resonance, vascular ultrasound and olfactory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged between 45 and 75 years
2. Spanish and/or Catalan speakers
3. Agreement with the study procedures and tests:

   1. Clinical Interview and questionnaires associated to risk factors
   2. Cognitive tests
   3. Blood sample extraction for DNA analysis
4. Close relative involvement for functional evaluation of the volunteer
5. Signature of informed consent

Exclusion Criteria:

1. Cognitive impairment: MMSE <26, o MIS <6, or orientation subtest of the Barcelona Test II <68, o category fluency (animals) <12
2. Functional status impairment: CDR > 0
3. Severe auditory and/or visual impairment
4. Neurodevelopmental and/or psychomotor disorder
5. Significant diseases that could currently interfere with cognition: renal failure on hemodialysis, liver cirrhosis, chronic lung disease with oxygen therapy, solid organ transplantation, fibromyalgia, active cancer in treatment or any other disease the investigator considers could affect the participant cognition
6. Major psychiatric disorders (DSM-IV-TR) or diseases that could affect cognitive abilities: major depression, bipolar disorder, schizophrenia and dementia.
7. Neurological disorders: Parkinson's disease, stroke, epilepsy and treatment with frequent seizures (> 1/month) in the past year, multiple sclerosis or other serious neurological disease.
8. Brain injury interfering with cognition: history of head trauma with parenchymal lesion or extraaxial macroscopic large vessel ischemic stroke or hemorrhagic stroke, brain surgery, brain tumors and other causes that can generate acquired brain damage (cerebral chemotherapy or radiotherapy)
9. Family history of Alzheimer's disease with autosomal dominant (3 affected in two different generations) and early onset age (<60 years).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cognitive normal men and woman aged 45-75 years
Sampling Method: Non-Probability Sample
Enrollment: 2743 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Factors influencing the cognitive performance through demanding tests of episodic memory and executive function | single Visit (up to 3 hours)
  The following tests will be administered:
  Verbal episodic memory: MBT (Memory Binding Test)
  WAIS-IV subsets: 1 Perceptual reasoning (Visual Puzzles) 2 Logical reasoning (Matrix Reasoning) 3 Executive attention and working memory (Digit span) 4 Speed of processing (Coding) 5 Abstract verbal reasoning (Similarities)
  Factors to be considered:
  Hypertension, diabetes mellitus, and metabolic syndrome APOE4 Cognitive reserve (including bilingualism) Pollution, exposure to toxics, diet
Culturally adapted validation in Spanish and Catalan of the MBT and determination of normative data for the population under study. | single visit (up to 3 hours)

SECONDARY OUTCOMES:
Assessment of the equivalence of the in person and over the phone administration to the close relative of the Clinical Dementia Rating (CDR). | single visit/telephone conversation (up to 10 min)
Genetic features of the population | 8 months after study start
  APOE genotyping is being performed
Identification of genetic determinants of neuroimaging phenotypes associated to Alzheimer's disease. | 5 years and 8 months after study start
  Brain MR (magnetic resonance) as well as GWAS (genome-wide association studies) are being performed
Assessment of the relationship between olfactory and cognitive performance | 5 years and 8 months after study start
  Olfaction is assessed with the Burghart Medical Technology (Wedel, Germany) kit containing 16 sniffing sticks
Analysis of the relationship between subclinical atherosclerosis and brain changes, cognitive performance and APOE genotype | 6 years and 8 months after study start
  Vascular ultrasound of femoral and carotid arteries will be performed

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Molinuevo, MD, PhD, Principal Investigator — Barcelonabeta Brain Research Center, Pasqual Maragall Foundation
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Spain

REFERENCES:
- [Derived] Cumplido-Mayoral I, Garcia-Prat M, Operto G, Falcon C, Shekari M, Cacciaglia R, Mila-Aloma M, Lorenzini L, Ingala S, Meije Wink A, Mutsaerts HJMM, Minguillon C, Fauria K, Molinuevo JL, Haller S, Chetelat G, Waldman A, Schwarz AJ, Barkhof F, Suridjan I, Kollmorgen G, Bayfield A, Zetterberg H, Blennow K, Suarez-Calvet M, Vilaplana V, Gispert JD; ALFA study; EPAD study; ADNI study; OASIS study. Biological brain age prediction using machine learning on structural neuroimaging data: Multi-cohort validation against biomarkers of Alzheimer's disease and neurodegeneration stratified by sex. Elife. 2023 Apr 17;12:e81067. doi: 10.7554/eLife.81067. PMID 37067031
- [Derived] Ciampa I, Operto G, Falcon C, Minguillon C, Castro de Moura M, Pineyro D, Esteller M, Molinuevo JL, Guigo R, Navarro A, Gispert JD, Vilor-Tejedor N, For The Alfa Study. Genetic Predisposition to Alzheimer's Disease Is Associated with Enlargement of Perivascular Spaces in Centrum Semiovale Region. Genes (Basel). 2021 May 27;12(6):825. doi: 10.3390/genes12060825. PMID 34072165
- [Derived] Sala-Vila A, Arenaza-Urquijo EM, Sanchez-Benavides G, Suarez-Calvet M, Mila-Aloma M, Grau-Rivera O, Gonzalez-de-Echavarri JM, Crous-Bou M, Minguillon C, Fauria K, Operto G, Falcon C, Salvado G, Cacciaglia R, Ingala S, Barkhof F, Schroder H, Scarmeas N, Gispert JD, Molinuevo JL; ALFA study. DHA intake relates to better cerebrovascular and neurodegeneration neuroimaging phenotypes in middle-aged adults at increased genetic risk of Alzheimer disease. Am J Clin Nutr. 2021 Jun 1;113(6):1627-1635. doi: 10.1093/ajcn/nqab016. PMID 33733657
- [Derived] Grau-Rivera O, Navalpotro-Gomez I, Sanchez-Benavides G, Suarez-Calvet M, Mila-Aloma M, Arenaza-Urquijo EM, Salvado G, Sala-Vila A, Shekari M, Gonzalez-de-Echavarri JM, Minguillon C, Ninerola-Baizan A, Perissinotti A, Simon M, Kollmorgen G, Zetterberg H, Blennow K, Gispert JD, Molinuevo JL; ALFA Study. Association of weight change with cerebrospinal fluid biomarkers and amyloid positron emission tomography in preclinical Alzheimer's disease. Alzheimers Res Ther. 2021 Feb 17;13(1):46. doi: 10.1186/s13195-021-00781-z. PMID 33597012
- [Derived] Vilor-Tejedor N, Operto G, Evans TE, Falcon C, Crous-Bou M, Minguillon C, Cacciaglia R, Mila-Aloma M, Grau-Rivera O, Suarez-Calvet M, Garrido-Martin D, Moran S, Esteller M, Adams HH, Molinuevo JL, Guigo R, Gispert JD; ALFA Study. Effect of BDNF Val66Met on hippocampal subfields volumes and compensatory interaction with APOE-epsilon4 in middle-age cognitively unimpaired individuals from the ALFA study. Brain Struct Funct. 2020 Nov;225(8):2331-2345. doi: 10.1007/s00429-020-02125-3. Epub 2020 Aug 17. PMID 32804326
- [Derived] Ingala S, Mazzai L, Sudre CH, Salvado G, Brugulat-Serrat A, Wottschel V, Falcon C, Operto G, Tijms B, Gispert JD, Molinuevo JL, Barkhof F; ALFA Study. The relation between APOE genotype and cerebral microbleeds in cognitively unimpaired middle- and old-aged individuals. Neurobiol Aging. 2020 Nov;95:104-114. doi: 10.1016/j.neurobiolaging.2020.06.015. Epub 2020 Jun 29. PMID 32791423